CLINICAL TRIAL: NCT03680742
Title: Contour Neurovascular System - European Pre-Market Unruptured Aneurysm Study (CERUS)
Brief Title: Contour Neurovascular System - European Pre-Market Unruptured Aneurysm
Acronym: CERUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cerus Endovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNX-099.D
Record Dates: First submitted 2018-09-18; First posted 2018-09-21 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated (Experimental): All eligible patients who underwent an attempt with the Contour device.
  Interventions: Device: Contour Neurovascular System

INTERVENTIONS:
Device: Contour Neurovascular System — The Contour Neurovascular System™ is an intrasaccular, self-expanding, embolization device intended for the treatment of unruptured intracranial aneurysms.

SUMMARY:
Cerus Endovascular is sponsoring a prospective, multi-center trial to document the safety and performance of the Contour Neurovascular System™ ("Contour").

The purpose of the study is to document safety and performance of the Contour in treatment for patients with intracranial aneurysms (IA). The data from the study will be reported as a Pre-Market study to the Notified Body to support CE Mark approval.

DETAILED DESCRIPTION:
Contour Neurovascular System™ European Pre-Market Unruptured Aneurysm Study (CERUS) initiated enrollment in October 2018 to assess the safety and effectiveness of the Contour Neurovascular System ("Contour") in treatment of intracranial aneurysms (IA) with the intended indication for endovascular embolization of saccular IA. This prospective, single-arm, multicenter study was conducted to document the safety and performance of the Contour in treatment for patients with an IA.

ELIGIBILITY:
Patients of all genders who meet all indications and contraindications will proceed to implantation.

Inclusion criteria

1. Patient's indication for treatment of unruptured aneurysm is according to the national/international guidelines.
2. Age 18-80 years at screening
3. Patients who are suitable for non-emergency endovascular embolization of saccular IAs
4. IA located at a bifurcation in the anterior or posterior circulation with dimensions consistent with implant size selection guidelines included in the IFU
5. Patient has the necessary mental capacity to participate and is willing and able to participate in the study for the duration of the study follow-up and is able to comply with study requirements
6. Patient able to able to give their informed consent can be included in this study. This must be demonstrated by means of a personally signed and dated informed consent document indicating that the subject has been informed of and understood all pertinent aspects of the study.

Exclusion criteria

The presence of condition that may create unacceptable risk during the aneurysm embolization procedure, such as patients with:

1. Ruptured aneurysm
2. Patient anatomy or physiology considered unsuitable for endovascular treatment
3. Contraindication for arterial access
4. Largest measured IA equatorial diameter >8.5 mm or <2 mm
5. Largest measured IA neck diameter >8 mm or <2 mm
6. Target IA contains other devices/implants (e.g., coils)
7. Known allergy to platinum, nickel or titanium
8. Known allergy to contrast agents
9. Contraindication to anticoagulants or platelet inhibitor medication
10. Stenosis of the target IA's parent vessel >50%
11. Anticoagulation medications such as warfarin that cannot be discontinued
12. Pregnant, breastfeeding or planning pregnancy in the next 2 years
13. Acute / chronic renal failure (including dialysis); Creatinine > 2.00 mg/dl or > 182 μmol/L
14. Myocardial Infarction, Stroke or TIA within the last 6 months
15. Any other medical issue within the brain that precludes the device implantation such as brain surgery, radiation in the target area of intervention, acute traumatic craniocerebral injury, etc.
16. Other medical conditions that cause an inability to comply with study requirements and/or that could increase the risk of neurovascular procedures or death within 2 years (e.g., liver failure, cancer, heart failure, chronic obstructive pulmonary disease, immunosuppression, neural disease, and hematologic disorders etc.)
17. Participating in another study with investigational devices or drugs that would confound the effects of the study outcomes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Liebig, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (6):
- Christian-Doppler-Klinik, Salzburg, Austria
- Odense University Hospital, Odense, Denmark
- Germany (4):
  - Klinikum Augsburg, Augsburg
  - UKSH Campus Kiel, Kiel
  - UKSH Campus Luebeck, Lübeck
  - Klinikum der Universitat München, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liebig T, Killer-Oberpfalzer M, Gal G, Schramm P, Berlis A, Dorn F, Jansen O, Fiehler J, Wodarg F. The Safety and Effectiveness of the Contour Neurovascular System (Contour) for the Treatment of Bifurcation Aneurysms: The CERUS Study. Neurosurgery. 2022 Mar 1;90(3):270-277. doi: 10.1227/NEU.0000000000001783. Epub 2021 Dec 29. PMID 35113830

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treated
Started | 34
Completed | 32
Not Completed | 2
Not completed — Unsuccessful Implant Attempt | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treated
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 6
  Denmark | 6
  Germany | 22

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: Percentage of Participants With Death of Any Non-accidental Cause or Major Disabling Stroke Within First 30 Days After Treatment or Major Disabling Stroke or Death Due to Neurological Cause From Day 31 to 6 Months After Treatment.
Description: The Primary Safety Endpoint is the percentage of subjects with death of any non-accidental cause or any major disabling stroke within the first 30 days after treatment or major disabling stroke or death due to neurological cause from day 31 to 6 months after treatment. Major Disabling Stroke is defined as an episode of neurological signs or symptoms that persist beyond 24 hours accompanied with evidence of ischemia/infarction on imaging that results in an increase of NIHSS from baseline by >= 4 points and/or an increase from mRS baseline by >2. An independent Clinical Events Committee adjudicated all data used for safety endpoint analyses.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 34
Participants | 1

2. Primary Outcome: Primary Performance Endpoint: Percentage of Subjects With Complete Aneurysm Occlusion at 6 Months.
Description: The Primary Performance Endpoint was the percentage of subjects with complete aneurysm occlusion at 6 months as adjudicated by an independent core laboratory. Occlusion was assessed using the Raymond-Roy occlusion scale (Class 1 - Complete occlusion; Class 2 - Residual neck; Class 3 - Residual aneurysm).
Time Frame: 6 months
Population: Subjects with 6-month cerebral angiograms assessed by the core laboratory.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 29
Participants
  Class 1 | 14
  Class 2 | 9
  Class 3 | 6

ADVERSE EVENTS:
Time Frame: 1 year (32 subjects); 1 month (2 subjects)
Arm/Group | Treated
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 13/34
Other Adverse Events (participants affected / at risk) | 9/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated (N=34)
Seizure (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 8 (10)
Thrombus (Nervous system disorders) | 1 (1)
Other - Procedure related (General disorders) | 5 (5)
Other - Not related to device or procedure (General disorders) | 3 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated (N=34)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Other - Not related to device or procedure (General disorders) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT03680742/Prot_001.pdf
  • Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT03680742/SAP_002.pdf